CLINICAL TRIAL: NCT05440487
Title: A Prospective Non-interventional Study to Assess Iron Chelation Therapy in Patients With Chronic Iron Overload
Brief Title: Study to Assess Iron Chelation Therapy in Patients With Chronic Iron Overload
Acronym: EXCALIBUR
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CICL670ADE14
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Chronic Iron Overload
Keywords: chronic iron overload; Germany; NIS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Iron chelator: Patients prescribed with Iron Chelators
  Interventions: Other: Iron chelator

INTERVENTIONS:
Other: Iron chelator — There is no treatment allocation. Patients administered approved Iron chelators by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This is a prospective, multicenter, non-interventional study. Findings are analyzed using epidemiological methods.

DETAILED DESCRIPTION:
This NIS shall document the therapy of chronic iron overload in a broad patient population with either of the approved iron chelators in Germany. The choice of patients and the therapy according to the SmPC follows the clinical routine exclusively. The regular observation time per patient is 24 months.

Corresponding to the clinical routine, follow up visits can be documented after approximately 1, 3, 6, 9, 12 and 18 month with a close out visit after 24 month. In case the iron chelator is switched, the visit scheme should be passed through once again.

ELIGIBILITY:
Inclusion Criteria:

Male and female adult patients suffering from chronic iron overload

* who never received an iron chelator directly before starting an iron chelation therapy
* who received an iron chelation therapy for less than 6 month
* who interrupted an iron chelation therapy for longer than 6 months and will receive an iron chelation therapy again
* who signed the informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult patients suffering from chronic iron overload receiving an iron chelation therapy
Sampling Method: Non-Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Efficiency of iron overload therapy | Up to 24 months
  Efficiency of iron chelation therapy is evaluated by the change of serum ferritin

SECONDARY OUTCOMES:
Number of patients treated with different iron chelators | Up to 24 months
  Number of patients treated with one of the three iron chelators approved in Germany.
Number of patients with therapy switch | Up to 24 months
  Number of patients with therapy switch in the standard clinical routine and the reason for the switch.
  The documentation of a therapy change is limited to the end of recruitment time (10/31/2019). From that date, the documentation of a change in therapy is no longer applicable.
Number of patients with dose adjustments | Up to 24 months
  Number of patients with dose adjustments during the observational period are collected
Number of patients with myelodyplastic syndromes or myeloproliferative neoplasms experiencing a hematologic response during an iron chelation therapy | Up to 24 months
  The analysis of a hematological response to iron chelation therapy should follow the effective criteria of the international working group
Number of patients with AEs and SAE | Up to 24 months
  Number of patients with Adverse Events and Serious Adverse Events is collected
Number of patients with side effects | Up to 24 months
  Side effects are defined as all adverse events, which are suspected to have a causality with the respective iron chelator.
  All events are reported in the eCRF and causality with iron chelator treatment is requested.
Treatment Satisfaction Questionnaire to Medication (TSQM) 1.4 | Up to 24 months
  TSQM is used to measure the Patients' self-reported satisfaction or dissatisfaction with the study treatment. The TSQM version 1.4 domain scores range from 0 to 100 with higher scores representing a higher satisfaction on that domain.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (91):
- Germany (91):
  - Novartis Investigative Site, Heidenheim, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Winnenden, Baden-Wurttemberg
  - Novartis Investigative Site, Aschaffenburg, Bavaria
  - Novartis Investigative Site, Bamberg, Bavaria
  - Novartis Investigative Site, Bayreuth, Bavaria
  - Novartis Investigative Site, Landshut, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Garbsen, Lower Saxony
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dortmund, North Rhine-Westphalia
  - Novartis Investigative Site, Duisburg, North Rhine-Westphalia
  - Novartis Investigative Site, Gelsenkirchen, North Rhine-Westphalia
  - Novartis Investigative Site, Iserlohn, Northrhine Westfalia
  - Novartis Investigative Site, Remscheid Innen, Northrhine Westfalia
  - Novartis Investigative Site, Neuwied, Rhineland-Palatinate
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Pirna, Saxony
  - Novartis Investigative Site, Zittau, Saxony
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Erfurt, Thuringia
  - Novartis Investigative Site, Altenburg
  - Novartis Investigative Site, Bad Liebenwerda
  - Novartis Investigative Site, Bad Mergentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Biberach
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Bremerhaven
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Donauwörth
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamelin
  - Novartis Investigative Site, Hamm
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Herrsching am Ammersee
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Hof
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Kronach
  - Novartis Investigative Site, Lemgo
  - Novartis Investigative Site, Lüdenscheid
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Naunhof
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Neustadt
  - Novartis Investigative Site, Nordhorn
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Passau
  - Novartis Investigative Site, Porta Westfalica
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rötha
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Schorndorf
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Speyer
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stolberg
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Traunstein
  - Novartis Investigative Site, Weiden
  - Novartis Investigative Site, Wesel
  - Novartis Investigative Site, Westerstede
  - Novartis Investigative Site, Wittenberg
  - Novartis Investigative Site, Wolfsburg
  - Novartis Investigative Site, Würselen
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CICL670ADE14 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17984